CLINICAL TRIAL: NCT05769972
Title: Randomized, Single-blind Clinical Trial to Evaluate the Efficacy of Cognitive Rehabilitation Using Inmersive Virtual Reality and Computer-based Cognitive Stimulation Versus Music Therapy on Cognitive Impairment Associated With Movement Disorders
Brief Title: Efficacy of Cognitive Rehabilitation Using Virtual Reality and Computer-based Cognitive Stimulation on Cognitive Impairment Associated to Movement Disorders
Acronym: CogMusT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-MOV-2021-28
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease; Huntington Disease
Keywords: Cognitive impairment; Cognitive rehabilitation; Virtual reality; Music therapy; Computer-based cognitive rehabilitation
MeSH Terms: conditions — Parkinson Disease; Huntington Disease; Cognitive Dysfunction | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Two interventions or each disease:
  Parkinson's disease:
Who Masked: Outcomes Assessor
Masking Description: Single-blind: outcomes assessor do not know where the participants are allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immersive Virtual Reality (Parkinson's disease) (Experimental)
  Interventions: Device: Immersive Virtual Reality (Parkinson's disease)
- Computer-based cognitive rehabilitation (Parkinson's disease) (Active Comparator)
  Interventions: Device: Computer-based cognitive rehabilitation (Parkinson's disease)
- Computer-based cognitive rehabilitation (Huntington's disease) (Experimental)
  Interventions: Device: Computer-based cognitive rehabilitation (Huntington's disease)
- Music-therapy (Huntington's disease) (Active Comparator)
  Interventions: Behavioral: Music-therapy (Huntington's disease)

INTERVENTIONS:
Device: Immersive Virtual Reality (Parkinson's disease) — This tool involves placing sensors in the space where it will be used, wearing virtual reality glasses, and using controllers to create realistic fictional spaces and interact with them. The program used for the study consists of an interface and a set of tasks designed specifically for the type of cognitive process deficits related to frontal function (executive functions) that are predominantly presented by patients with cognitive impairment associated with Parkinson's disease. This is due to the effect of the disease's pathophysiology on a series of brain circuits and structures that range from the basal ganglia to the frontal lobe. The affected functions correspond to the individual's ability to plan, sequence, organize, make decisions, be flexible, abstract, conceptualize, inhibit, among others.
  Arms: Immersive Virtual Reality (Parkinson's disease)
Device: Computer-based cognitive rehabilitation (Parkinson's disease) — This consists of a 24-week computerized cognitive stimulation program using the NeuronUp software. The intervention includes a limited number of tasks developed ad hoc by NeuronUp and the researchers specifically aimed at stimulating the cognitive domains typically affected in movement disorders. These are cognitive processes mostly ascribed to frontal function, as well as other less prevalent but equally disabling processes mainly associated with basal ganglia and fronto-striatal circuitry, such as executive functions, attention and working memory, language, processing speed, and social cognition. Thus, the programs are the same for PD and HD, although the parameters of the number of errors, level of difficulty, and number of correct answers required to advance to the next level have been adjusted to be more demanding in PD and less in HD, with the aim of customizing this type of intervention to the clinical characteristics of each disease.
  Arms: Computer-based cognitive rehabilitation (Parkinson's disease)
Device: Computer-based cognitive rehabilitation (Huntington's disease) — This consists of a 24-week computerized cognitive stimulation program using the NeuronUp software. The intervention includes a limited number of tasks developed ad hoc by NeuronUp and the researchers specifically aimed at stimulating the cognitive domains typically affected in movement disorders. These are cognitive processes mostly ascribed to frontal function, as well as other less prevalent but equally disabling processes mainly associated with basal ganglia and fronto-striatal circuitry, such as executive functions, attention and working memory, language, processing speed, and social cognition. Thus, the programs are the same for PD and HD, although the parameters of the number of errors, level of difficulty, and number of correct answers required to advance to the next level have been adjusted to be more demanding in PD and less in HD, with the aim of customizing this type of intervention to the clinical characteristics of each disease.
  Arms: Computer-based cognitive rehabilitation (Huntington's disease)
Behavioral: Music-therapy (Huntington's disease) — The process used in each session will be standardized, while the content will be flexible, administering the guidelines according to the mood of the patients and their needs at that time. The therapist's clinical experience will guide them, providing sufficient space for flexible adaptation within the treatment guideline. While the sessions will be standardized, without limiting the music therapist in their interactions, the intervention itself will be applied during the experimental period, using all of the cognitive music therapy exercises detailed below in all groups: auditive perception training, musical sensorial orientation, control of musical attention, training of musical executive function, training in musical mnemotecnia and associative training of mood and musical memory
  Arms: Music-therapy (Huntington's disease)

SUMMARY:
Mild cognitive impairment associated with movement disorders occurs in up to one third of patients in early stages of the disease, and confers an increased risk of developing dementia. Non-pharmacological interventions to improve cognition have so far been based on computer-based cognitive stimulation and rehabilitation programs. These interventions base their mechanism of action on neuroplasticity and how improvements in cognitive function will generalize to functional improvement.

Despite having shown certain indicators of efficacy in previous exploratory studies and clinical trials, cognitive rehabilitation continues to show insufficient evidence and requires further study.

To date, there are no previous studies using immersive virtual reality (IVR) to improve cognition. Both IVR and cognitive stimulation are based on the premise that they allow the simulation of ecological environments for rehabilitation than conventional rehabilitation, as well as being more efficient by allowing control of extraneous variables and providing safe spaces for patients. The only PD rehabilitation studies that have been conducted using IVR aimed to improve gait and balance disturbances compared to conventional physiotherapy treatment or non-immersive virtual reality (NIVR).

We hypothesize that a cognitive rehabilitation program using IVR or computer-mediated cognitive stimulation could have a greater beneficial effect on the cognitive status of patients with cognitive impairment associated with movement disorders compared to other modalities such as music therapy, delaying the worsening of cognitive functions.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by progressive neuronal loss in the substantia nigra of the midbrain, as well as in other areas such as the pons, diencephalon, limbic system, and temporal cortex, which is accompanied by the deposition of alpha-synuclein in surviving neurons. (1) This neurodegeneration clinically manifests as motor symptoms (bradykinesia, rigidity, tremor) and non-motor symptoms (depression, anxiety, apathy, and cognitive impairment, among others).

Cognitive impairment associated with PD is currently recognized as one of the most relevant non-motor symptoms due to the significant impact it has on families and the economic cost it represents for public health. Dementia associated with PD is invariably preceded by a phase of mild cognitive impairment (MCI), characterized by the presence of alteration in neuropsychological tests without significant impact on the patient's functional capacity. Patients with MCI have a higher risk of developing dementia during the course of the disease. Specifically, conversion rates of 27.8% in the first year and up to 45.5% after 3 years have been described. (2)

Cognitive impairment associated with PD depends both on dopaminergic denervation of the nigrostriatal circuit (and secondary failure of fronto-subcortical circuits) and on the involvement of cholinergic brainstem structures, which project widely in the brain. (3) There is also growing evidence that cognitive impairment in PD is not only related to the deposition of alpha-synuclein, but that the deposition of beta-amyloid (characteristic of Alzheimer's disease) also plays an important role. (4)

Huntington's disease (HD) is a dominant autosomal neurodegenerative disease caused by an expansion of CAG in exon 1 of the gene that encodes for huntingtin on chromosome 4. This abnormal expansion of CAG gives rise to mutant huntingtin, considered the main protein involved in the pathophysiology of HD. (5) Individuals who carry the mutation and have ≥40 CAG repeats will inevitably show progressive motor (chorea, bradykinesia, and dystonia), cognitive (cognitive impairment and dementia), psychiatric (depression, apathy, perseverative behavior, irritability, among others), and functional deterioration in adulthood. The average age of onset of motor symptoms is around 45 years, and the course of the disease is approximately 10-20 years. (6)

Cognitive impairment associated with HD has been mainly attributed to progressive atrophy of the basal ganglia together with the disruption of fronto-subcortical circuits that accompany it. However, other diffuse brain changes, including alterations in cerebral white matter and posterior cortical atrophy, have also been shown to contribute to cognitive impairment. (7, 8)

The treatments currently available are basically symptomatic, and so far no drug has been found to alter the natural history of these diseases. (9) Finding a new target or treatment to reduce the progressive nature of the disease represents an important challenge from a scientific, healthcare, and social perspective. Specifically, acting effectively in the early stages of cognitive impairment in PD and HD to reduce the conversion rate to dementia would represent an immeasurable benefit.

The goal of cognitive rehabilitation is to improve a person's functional performance and compensate for cognitive deficits resulting from brain damage in order to reduce functional limitations, increasing people's ability to perform daily activities. (10) The ultimate purpose is to improve the quality of life of people. (11, 12)

Cognitive functions are interrelated and interdependent at an anatomical level when functional responses are required. They involve multiple types and levels of processing. When an external or internal activity is carried out, neuronal networks are combined, either modularly or through large-scale networks. These combinations recruit specific neuropsychological processes that are carried out for execution. From visual recognition to initiation processes of behavior (automatic or not), impulse control, or the development of metacognitive strategies that plan behavior. Therefore, from an applied point of view, formulating rehabilitation activities that cover the entire range of processes, discretely but also holistically, would be the appropriate way of application to achieve therapy that is as ecologically, customizable, and generalizable as possible.

The mechanism of action on which cognitive rehabilitation or stimulation programs are based is neuroplasticity. This is defined as the brain's ability to reorganize its patterns of neuronal connectivity by generating new synapses, adjusting its functionality. Neuroplasticity is present both in normal aging and in conditions of acquired brain damage or dementias. The greater efficacy of these types of programs has been found in patients with acquired brain damage (stroke, traumatic brain injury, among others) and to a lesser extent in the field of dementias, although it has shown some benefit compared to usual treatment. Today there is no established consensus regarding the effect that occurs by taking advantage of the plasticity phenomenon, as it depends on multiple factors: type of deterioration, age, recovery process, cognitive reserve, genetic factors, among others.

Plasticity can improve learning processes at three levels: a neuronal level, a synaptic level, and a network level (changes in functional connectivity). These levels are not mutually exclusive. The remodeling of short- and long-term neuronal activity patterns, including the formation, elimination, and change in firing frequencies and thresholds, as well as the sprouting of new axons, are the main ways to achieve neuronal organization through experience and maturation. Neurotrophic factors are also modified by experience through epigenetic regulation.

The effect that music therapy has on rhythm and its relationship to the motor aspects of the basal ganglia suggests that music therapy could be useful in the field of emotional complications of neurodegenerative diseases. Studies on music therapy in Parkinson's disease have shown efficacy and usefulness as therapy for speech rehabilitation or improvement of gait, posture, and balance. Since music therapy is not associated with significant adverse effects, music appears as a viable and attractive option as an active control treatment.

Conclusions:

Cognitive impairment associated with movement disorders has a significant negative impact on the autonomy and quality of life of both patients and families and makes them highly dependent on healthcare and social resources. The treatments currently available are basically symptomatic, and so far no therapy has been found to change the natural history of these diseases.

The lack of pharmacological strategies to stop or slow down cognitive decline associated with neurodegenerative diseases, specifically movement disorders, highlights the importance of developing non-pharmacological therapeutic strategies to change the course of cognitive decline and achieve greater functionality. Cognitive stimulation programs based on RVI or RVNI have the characteristic of creating ecologically valid environments that allow for practice based on the interaction of different cognitive processes depending on the task, and ultimately allow for generalization in daily life through learning and automation of routines or optimization of neural networks, generation of new synapses, and changes in neuronal firing that allow for neuroplasticity.

So far, evidence on cognitive rehabilitation in the field of movement disorders is based on cognitive stimulation studies involving the repetition of tasks focused on one or more cognitive processes without clear ecological validity, or in studies based on virtual reality that are limited to improving motor function in Parkinson's disease (24, 25, 26, 27, 28). To date, the heterogeneity in the conceptualization of cognitive decline in movement disorders without following consensus criteria for including patients in clinical trials has led to demonstrating limited efficacy or non-comparability with other studies. The importance of correctly classifying patients based on their cognitive status is crucial for the proper design of trials aimed at improving cognitive function in movement disorders (7, 26, 29, 30).

Therefore, we have designed a study focused on evaluating the effect of cognitive rehabilitation based on RVI and computer-based cognitive stimulation on cognitive decline in movement disorders. Given the natural history of these types of diseases, we have the possibility of detecting cognitive changes in a relatively short period of time using appropriate tools (31, 32). The PD-CRS has been shown to be capable of detecting changes in cognitive status in Parkinson's disease and Huntington's disease over time (good sensitivity to change), being able to detect clinically relevant differences in a period of 6 months. To assess clinical relevance, the Clinical Global Impression of Change scale was used, with a change of 11-14 points in the PD-CRS being the minimum to consider that there is a clinical impact. For this reason, we consider that a single-blind clinical trial of 6 months duration would be sufficient to demonstrate significant differences between the cognitive performance of the control group (music therapy) and the RVI or computer-based cognitive stimulation group.

ELIGIBILITY:
Inclusion Criteria:

* Patient capable of understanding, signing and dating the written informed consent at baseline visit prior to randomization.
* Patient diagnosed with Parkinson's disease (Movement Disorder Society PD Criteria) or Huntington's disease.
* Patient with Hoehn and Yahr stage I-III for PD, and Shoulson and Fahn stage I-II for HD.
* Patient with a score on the Parkinson's Disease Cognitive Rating Scale (PD-CRS) >83, who present subjective memory complaints will be included in "group I: subjective memory complaints".
* Patient with a score on the Parkinson's Disease Cognitive Rating Scale (PD-CRS) between 64 and 83, both inclusive, will be included in "group II: mild cognitive impairment".
* Patient diagnosed with Parkinson's disease with stable dopaminergic treatment in the last 4 weeks.
* Patient capable and willing to comply with study visits as detailed in the protocol.

Exclusion Criteria:

* Illiterate patients.
* Patients with severe vision or hearing impairment.
* History of deep brain stimulation surgery.
* Patients diagnosed with severe dementia (possible or probable) associated with Parkinson's disease, according to the Clinical Diagnostic Criteria for Dementia Associated with PD with a score of >2 on the CRD or with Huntington's disease.
* Patients with active psychosis in the form of incapacitating delusional ideation.
* Patients who were under experimental treatment in the 2 months prior to the selection period.
* Patients with any of the following conditions:
* Life expectancy of less than 6 months.
* Any severe or uncontrolled medical condition.
* Patients with a history of poor treatment compliance or drug/alcohol abuse that may interfere with the patient's ability to comply with the study protocol or give informed consent.
* Pregnancy or breastfeeding.
* Contraindications for MRI*.

  * Except for patients with Parkinson's disease (PD), since MRI is optional for these patients. Therefore, if there are contraindications for MRI, they can still participate without undergoing MRI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease - Cognitive Rating Scale (PD-CRS) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Background] Lang AE, Lozano AM. Parkinson's disease. First of two parts. N Engl J Med. 1998 Oct 8;339(15):1044-53. doi: 10.1056/NEJM199810083391506. No abstract available. PMID 9761807
- [Background] Pedersen KF, Larsen JP, Tysnes OB, Alves G. Prognosis of mild cognitive impairment in early Parkinson disease: the Norwegian ParkWest study. JAMA Neurol. 2013 May;70(5):580-6. doi: 10.1001/jamaneurol.2013.2110. PMID 23529397
- [Background] Pavese N, Rivero-Bosch M, Lewis SJ, Whone AL, Brooks DJ. Progression of monoaminergic dysfunction in Parkinson's disease: a longitudinal 18F-dopa PET study. Neuroimage. 2011 Jun 1;56(3):1463-8. doi: 10.1016/j.neuroimage.2011.03.012. Epub 2011 Mar 17. PMID 21396455
- [Background] Clinton LK, Blurton-Jones M, Myczek K, Trojanowski JQ, LaFerla FM. Synergistic Interactions between Abeta, tau, and alpha-synuclein: acceleration of neuropathology and cognitive decline. J Neurosci. 2010 May 26;30(21):7281-9. doi: 10.1523/JNEUROSCI.0490-10.2010. PMID 20505094
- [Background] Walker FO. Huntington's disease. Lancet. 2007 Jan 20;369(9557):218-28. doi: 10.1016/S0140-6736(07)60111-1. PMID 17240289
- [Background] Sorensen SA, Fenger K. Causes of death in patients with Huntington's disease and in unaffected first degree relatives. J Med Genet. 1992 Dec;29(12):911-4. doi: 10.1136/jmg.29.12.911. PMID 1479606
- [Background] Peavy GM, Jacobson MW, Goldstein JL, Hamilton JM, Kane A, Gamst AC, Lessig SL, Lee JC, Corey-Bloom J. Cognitive and functional decline in Huntington's disease: dementia criteria revisited. Mov Disord. 2010 Jul 15;25(9):1163-9. doi: 10.1002/mds.22953. PMID 20629124
- [Background] Sampedro F, Martinez-Horta S, Perez-Perez J, Horta-Barba A, Lopez-Mora DA, Camacho V, Fernandez-Leon A, Gomez-Anson B, Carrio I, Kulisevsky J. Cortical atrophic-hypometabolic dissociation in the transition from premanifest to early-stage Huntington's disease. Eur J Nucl Med Mol Imaging. 2019 May;46(5):1111-1116. doi: 10.1007/s00259-018-4257-z. Epub 2019 Jan 9. PMID 30627816
- [Background] Harikrishna Reddy D, Misra S, Medhi B. Advances in drug development for Parkinson's disease: present status. Pharmacology. 2014;93(5-6):260-71. doi: 10.1159/000362419. Epub 2014 Aug 1. PMID 25096413
- [Background] Oberholzer M, Muri RM. Neurorehabilitation of Traumatic Brain Injury (TBI): A Clinical Review. Med Sci (Basel). 2019 Mar 18;7(3):47. doi: 10.3390/medsci7030047. PMID 30889900
- [Background] Prigatano GP, Fordyce DJ, Zeiner HK, Roueche JR, Pepping M, Wood BC. Neuropsychological rehabilitation after closed head injury in young adults. J Neurol Neurosurg Psychiatry. 1984 May;47(5):505-13. doi: 10.1136/jnnp.47.5.505. PMID 6736983
- [Background] Sohlberg MM, Mateer CA. Introduction to cognitive rehabilitation: Theory and practice. Guilford Press. 1989
- [Background] Cicerone KD, Goldin Y, Ganci K, Rosenbaum A, Wethe JV, Langenbahn DM, Malec JF, Bergquist TF, Kingsley K, Nagele D, Trexler L, Fraas M, Bogdanova Y, Harley JP. Evidence-Based Cognitive Rehabilitation: Systematic Review of the Literature From 2009 Through 2014. Arch Phys Med Rehabil. 2019 Aug;100(8):1515-1533. doi: 10.1016/j.apmr.2019.02.011. Epub 2019 Mar 26. PMID 30926291
- [Background] Orgeta V, McDonald KR, Poliakoff E, Hindle JV, Clare L, Leroi I. Cognitive training interventions for dementia and mild cognitive impairment in Parkinson's disease. Cochrane Database Syst Rev. 2020 Feb 26;2(2):CD011961. doi: 10.1002/14651858.CD011961.pub2. PMID 32101639
- [Background] Bahar-Fuchs A, Martyr A, Goh AM, Sabates J, Clare L. Cognitive training for people with mild to moderate dementia. Cochrane Database Syst Rev. 2019 Mar 25;3(3):CD013069. doi: 10.1002/14651858.CD013069.pub2. PMID 30909318
- [Background] Fernandez Lopez R, Antoli A. Computer-based cognitive interventions in acquired brain injury: A systematic review and meta-analysis of randomized controlled trials. PLoS One. 2020 Jul 9;15(7):e0235510. doi: 10.1371/journal.pone.0235510. eCollection 2020. PMID 32645046
- [Background] Dobkin BH. Curiosity and cure: translational research strategies for neural repair-mediated rehabilitation. Dev Neurobiol. 2007 Aug;67(9):1133-47. doi: 10.1002/dneu.20514. PMID 17514711
- [Background] Berlucchi G. Brain plasticity and cognitive neurorehabilitation. Neuropsychol Rehabil. 2011 Oct;21(5):560-78. doi: 10.1080/09602011.2011.573255. Epub 2011 May 24. PMID 21563013
- [Background] Alvarez VA, Sabatini BL. Anatomical and physiological plasticity of dendritic spines. Annu Rev Neurosci. 2007;30:79-97. doi: 10.1146/annurev.neuro.30.051606.094222. PMID 17280523
- [Background] Bloem BR, de Vries NM, Ebersbach G. Nonpharmacological treatments for patients with Parkinson's disease. Mov Disord. 2015 Sep 15;30(11):1504-20. doi: 10.1002/mds.26363. Epub 2015 Aug 14. PMID 26274930
- [Background] Raglio A, Bellandi D, Baiardi P, Gianotti M, Ubezio MC, Zanacchi E, Granieri E, Imbriani M, Stramba-Badiale M. Effect of Active Music Therapy and Individualized Listening to Music on Dementia: A Multicenter Randomized Controlled Trial. J Am Geriatr Soc. 2015 Aug;63(8):1534-9. doi: 10.1111/jgs.13558. PMID 26289682
- [Background] Barnish J, Atkinson RA, Barran SM, Barnish MS. Potential Benefit of Singing for People with Parkinson's Disease: A Systematic Review. J Parkinsons Dis. 2016 Jun 3;6(3):473-84. doi: 10.3233/JPD-160837. PMID 27258698
- [Background] Martinez-Molina N, Mas-Herrero E, Rodriguez-Fornells A, Zatorre RJ, Marco-Pallares J. Neural correlates of specific musical anhedonia. Proc Natl Acad Sci U S A. 2016 Nov 15;113(46):E7337-E7345. doi: 10.1073/pnas.1611211113. Epub 2016 Oct 31. PMID 27799544
- [Background] Canning CG, Allen NE, Nackaerts E, Paul SS, Nieuwboer A, Gilat M. Virtual reality in research and rehabilitation of gait and balance in Parkinson disease. Nat Rev Neurol. 2020 Aug;16(8):409-425. doi: 10.1038/s41582-020-0370-2. Epub 2020 Jun 26. PMID 32591756
- [Background] Diez-Cirarda M, Ibarretxe-Bilbao N, Pena J, Ojeda N. Neurorehabilitation in Parkinson's Disease: A Critical Review of Cognitive Rehabilitation Effects on Cognition and Brain. Neural Plast. 2018 May 6;2018:2651918. doi: 10.1155/2018/2651918. eCollection 2018. PMID 29853840
- [Background] Biundo R, Weis L, Fiorenzato E, Antonini A. Cognitive Rehabilitation in Parkinson's Disease: Is it Feasible? Arch Clin Neuropsychol. 2017 Nov 1;32(7):840-860. doi: 10.1093/arclin/acx092. PMID 28961738
- [Background] Bartlett DM, Govus A, Rankin T, Lampit A, Feindel K, Poudel G, Teo WP, Lo J, Georgiou-Karistianis N, Ziman MR, Cruickshank TM. The effects of multidisciplinary rehabilitation on neuroimaging, biological, cognitive and motor outcomes in individuals with premanifest Huntington's disease. J Neurol Sci. 2020 Sep 15;416:117022. doi: 10.1016/j.jns.2020.117022. Epub 2020 Jul 12. PMID 32688143
- [Background] van Walsem MR, Piira A, Mikalsen G, Fossmo HL, Howe EI, Knutsen SF, Frich JC. Cognitive Performance After a One-Year Multidisciplinary Intensive Rehabilitation Program for Huntington's Disease: An Observational Study. J Huntingtons Dis. 2018;7(4):379-389. doi: 10.3233/JHD-180294. PMID 30320595
- [Background] Mestre TA, Bachoud-Levi AC, Marinus J, Stout JC, Paulsen JS, Como P, Duff K, Sampaio C, Goetz CG, Cubo E, Stebbins GT, Martinez-Martin P; Members of the MDS Committee on Rating Scales Development. Rating scales for cognition in Huntington's disease: Critique and recommendations. Mov Disord. 2018 Feb;33(2):187-195. doi: 10.1002/mds.27227. Epub 2017 Dec 26. PMID 29278291
- [Background] Litvan I, Goldman JG, Troster AI, Schmand BA, Weintraub D, Petersen RC, Mollenhauer B, Adler CH, Marder K, Williams-Gray CH, Aarsland D, Kulisevsky J, Rodriguez-Oroz MC, Burn DJ, Barker RA, Emre M. Diagnostic criteria for mild cognitive impairment in Parkinson's disease: Movement Disorder Society Task Force guidelines. Mov Disord. 2012 Mar;27(3):349-56. doi: 10.1002/mds.24893. Epub 2012 Jan 24. PMID 22275317
- [Background] Fernandez de Bobadilla R, Pagonabarraga J, Martinez-Horta S, Pascual-Sedano B, Campolongo A, Kulisevsky J. Parkinson's disease-cognitive rating scale: psychometrics for mild cognitive impairment. Mov Disord. 2013 Sep;28(10):1376-83. doi: 10.1002/mds.25568. Epub 2013 Jul 19. PMID 23873810
- [Background] Martinez-Horta S, Horta-Barba A, Perez-Perez J, Sampedro F, de Lucia N, De Michele G, Kehrer S, Priller J, Migliore S, Squitieri F, Castaldo A, Mariotti C, Mananes V, Lopez-Sendon JL, Rodriguez N, Martinez-Descals A, Garcia-Ruiz P, Julio F, Januario C, Delussi M, de Tommaso M, Noguera S, Ruiz-Idiago J, Sitek EJ, Nuzzi A, Pagonabarraga J, Kulisevsky J; Cognitive Phenotype Working Group of the European Huntington's Disease Network. Utility of the Parkinson's disease-Cognitive Rating Scale for the screening of global cognitive status in Huntington's disease. J Neurol. 2020 May;267(5):1527-1535. doi: 10.1007/s00415-020-09730-6. Epub 2020 Feb 7. PMID 32030521
- [Derived] Puig-Davi A, Moreu-Valls A, Aracil-Bolanos I, Fernandez-Cocano A, Rodriguez-Antiguedad J, Kulisevsky G, Horta-Barba A, Pagonabarraga J, Kulisevsky J, Martinez-Horta S. Effects of immersive virtual reality and adaptive cognitive training on cognition and function in parkinson's disease mild cognitive impairment: a randomized clinical trial. Sci Rep. 2026 Jan 25. doi: 10.1038/s41598-025-31833-1. Online ahead of print. PMID 41582160
- [Derived] Moreu-Valls A, Puig-Davi A, Martinez-Horta S, Kulisevsky G, Sampedro F, Perez-Perez J, Horta-Barba A, Olmedo-Saura G, Pagonabarraga J, Kulisevsky J. A randomized clinical trial to evaluate the efficacy of cognitive rehabilitation and music therapy in mild cognitive impairment in Huntington's disease. J Neurol. 2025 Feb 12;272(3):202. doi: 10.1007/s00415-025-12927-2. PMID 39934473